CLINICAL TRIAL: NCT07047768
Title: Artificial Intelligence for Respiratory Infections SEverity Prediction
Acronym: AIRISE
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_1114_1
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Infectious Respiratory Diseases; Hospitalized Patients; Adult Patients
Keywords: Prediction; Artificial Intelligence; Infectious respiratory diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with acute lower respiratory tract infections (ALRTI): Adult patients (aged ≥ 18 years) admitted to the emergency department and/or hospitalized in one of the Hospices Civils de Lyon departments for a respiratory infection between January 1, 2017, and April 30, 2024.
  Interventions: Other: No intervention : data-based study

INTERVENTIONS:
Other: No intervention : data-based study — No intervention : data-based study

SUMMARY:
Health Data Warehouses (HDWs) are a major resource for the development of artificial intelligence (AI) applied to predictive and personalized medicine. We propose a project leveraging the HDW of the Hospices Civils de Lyon (HCL) to study acute lower respiratory tract infections (ALRTIs), a major public health issue due to their impact on morbidity, mortality, and healthcare costs. The COVID-19 pandemic has further highlighted their burden and complexity.

ALRTIs can be caused by viral agents (e.g., influenza, RSV, SARS-CoV-2) or bacterial pathogens (e.g., pneumococcus, mycoplasma, legionella), and may be acquired in the community or during hospitalization. Given their frequency and potential severity, early identification of patients at risk of clinical deterioration is crucial, especially those likely to require intensive care.

The recent deployment of the HCL HDW now allows for the structured extraction, linkage, and storage of administrative, clinical, biological, and pharmaceutical data. This system supports the reconstruction of each patient's care trajectory and clinical history, offering new opportunities for advanced modeling.

In recent years, several predictive tools have been developed to estimate the severity or prognosis of respiratory infections, including PSI/FINE, qSOFA, CURB-65, the EPIC sepsis model, and early warning systems (EWS). The COVID-19 crisis spurred the creation of new scores and models to predict clinical outcomes or mortality, as well as online tools and apps for clinicians. However, many of these tools rely on limited datasets (often single-center or small cohorts), static variables (e.g., comorbidities), and do not consider the temporal dynamics of patient data.

Some research teams have explored the use of multicenter data and machine learning (e.g., MLHO-Machine Learning to predict Health Outcomes), notably to model COVID-19 outcomes. Nonetheless, most models lack integration of longitudinal clinical and biological data, and few are generalizable to all respiratory infections. Additionally, existing tools rarely account for real-time contextual variables such as current levels of population immunity or vaccine availability.

Our project aims to develop a dynamic AI-based detection algorithm to predict the risk of ICU admission in patients with ALRTIs. The model will be trained on retrospective HDW data from the HCL, including the evolution of vital signs, laboratory values, treatments, and demographic factors. By capturing temporal trends and clinical trajectories, our algorithm will go beyond static scoring systems and offer real-time risk stratification.

Ultimately, this algorithm could be embedded in hospital information systems as a clinical decision support tool. By generating alerts for early signs of deterioration, it would enable more timely interventions, resource optimization, and improved patient outcomes.

This approach differs from existing models in two fundamental ways. First, it covers a broad patient population with viral and bacterial pneumonia of both community and hospital origin. Second, it explicitly incorporates the longitudinal dimension of health data, allowing the model to learn from dynamic changes in patient condition. This temporal perspective is key to improving prediction accuracy and enabling early detection of deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥ 18 years);
* With a visit to the emergency department and/or hospitalization in one of the Hospices Civils de Lyon departments;
* With a diagnosis of lower respiratory tract infection (ICD-10 code);
* Between January 1, 2017, and April 30, 2024;
* Who did not object to participating in the study.

Exclusion Criteria:

* Patients under 18 years of age at the time of care;
* Patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged ≥ 18 years) admitted to the emergency department and/or hospitalized in one of the Hospices Civils de Lyon departments for a respiratory infection between January 1, 2017, and April 30, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 52000 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Admission to intensive care unit | Adult patients (aged ≥ 18 years) admitted to the emergency department and/or hospitalized in one of the Hospices Civils de Lyon departments for a respiratory infection between January 1, 2017, and April 30, 2024.
  The primary outcome was admission to intensive care unit during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Hygiène, épidémiologie, infectiovigilance et prévention GHN, Hôpital Croix-Rousse, Lyon, France